CLINICAL TRIAL: NCT00929071
Title: Safety and Efficacy of the Addition of 0.3% Lidocaine With EVOLENCE®
Acronym: AD-1016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weinkle, Susan H., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS DP101L - US - 02
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Aging; Pain
Keywords: wrinkles; dermal filler; collagen; soft tissue augmentation; lidocaine; aesthetic
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain assessment for Evolence/topical anesthetic (Experimental): Assess injection pain severity for a one time 1.0 mL injection of Evolence with 0.2 ml of topical anesthetic, applied 30 minutes prior to injection, to the left nasolabial fold of each participant .
  Interventions: Device: Evolence; Drug: topical anesthetic
- Pain assessment for Evolence/Lidocaine (Experimental): Assess injection pain severity for a one time 1.0 mL injection of Evolence mixed with 0.18 mL of 2% lidocaine (0.3% final lidocaine-HCl) in the right nasolabial fold of each participant.
  Interventions: Device: Evolence; Device: Lidocaine

INTERVENTIONS:
Device: Evolence — Injectable collagen
  Other Names: collagen; Dermicol-P35 27G
Device: Lidocaine — admix anesthetic
  Arms: Pain assessment for Evolence/Lidocaine
Drug: topical anesthetic
  Arms: Pain assessment for Evolence/topical anesthetic

SUMMARY:
The study doctor will give EVOLENCE® mixed with Lidocaine to people in this study to see if it effectively reduces pain while injecting and works to correct nasolabial wrinkles.

The product being used in this study is EVOLENCE®, which is currently marketed in the United States for the cosmetic correction of soft tissue contour deficiencies (including wrinkles), and been approved by the U.S. Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The aim of this study is to determine if the admixture of lidocaine can effectively be used to mediate pain relief during the injection of EVOLENCE® while achieving cosmetic correction.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and voluntary signature (including date) of an informed consent document
* Healthy male or female > 18 years of age
* Clinical evidence of bilateral, fully visible aging defects in the nasolabial area with grades 2.0, 2.5, or 3.0 on the Modified Fitzpatrick Wrinkle Scale (MFWS section 6.5)
* Willingness to receive EVOLENCE® injections in areas of aging defects (wrinkles)
* Willingness and ability to comply with the requirements of this protocol

Exclusion Criteria:

* History of multiple severe allergies (food, drug, or substances) and/or anaphylactic shock
* Subjects with a history of a bleeding disorder, or receiving chronic anti-platelet therapy or other chronic anticoagulant medication
* Subject on low-dose aspirin therapy or a non-steroidal anti-inflammatory drug, not interrupted at least 10 days prior to injection and/or resumed within 1 week after injection
* History of allergies and/or sensitivity to porcine, bovine and human collagen, lidocaine, local anesthetics products or natural rubber latex
* Autoimmune or collagen vascular disease, or connective tissue disease
* Active skin disease, inflammation or related condition such as infection, psoriasis and herpes zoster near or on the nasolabial folds area at study entry and/or within 6 months prior to study entry
* Previous tissue augmentation - permanent implants or hyaluronic acid within 6 months or EVOLENCE® within 12 months in the treatment area
* Currently being treated with immunosuppressive drugs, chemotherapy agents or systemic steroids or has been treated within the last 3 months prior to study entry
* Botulinum-toxin A within 6 weeks in treatment area
* Received any investigational products within 30 days prior to the study enrollment
* Females of Childbearing Potential
* Any clinically significant organic disease or other medical condition that in the opinion of the PI, makes the subject a poor candidate for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Weinkle, MD, Principal Investigator — Private Practice
Locations (1):
- Susan Weinkle, Private Practice, Bradenton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Assess a difference in immediate post-injection pain of Evolence/topical anesthetic at the left nasolabial fold vs Evolence/Lidocaine at the right nasolabial fold.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pain Assessment: Assess injection pain of Evolence/topical anesthetic vs Evolence/Lidocaine mixture upon injection
Arm/Group | Pain Assessment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Immediate Post-injection Pain Severity by Subject
Description: Subjects assessment of immediate post-injection pain severity using a visual analogue scale (VAS) 100 mm in length, ranging from no pain (0) to unbearable pain (100).
Time Frame: immediate post-injection
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: nasolabial folds
Groups:
- Pain Assessment for Evolence/Topical Anesthetic: Assess injection pain of Evolence/topical anesthetic left nasolabial fold
  collagen: Injectable collagen
  topical anesthetic
- Pain Assessment for Evolence/Lidocaine: Assess injection pain of Evolence/Lidocaine right nasolabial fold
  collagen: Injectable collagen
  Lidocaine: admix anesthetic
Arm/Group | Pain Assessment for Evolence/Topical Anesthetic | Pain Assessment for Evolence/Lidocaine
Number analyzed (Participants) | 10 | 10
Number analyzed (nasolabial folds) | 10 | 10
units on a scale | 6.3 (2.0) | 2.0 (1.0)

2. Primary Outcome: Assessment of Immediate Post-injection Pain Severity by Investigator
Description: Investigators assessment of immediate post-injection pain severity using Thermometer Pain Scale (TPS) with a range of 0-10 where 0=no pain and 10=worst possible pain
Time Frame: immediate post injection
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: nasolabial folds
Groups:
- Pain Assessment for Evolence/Topical Anesthetic: Assess injection pain of Evolence/topical anesthetic
  collagen: Injectable collagen
  topical anesthetic
- Pain Assessment for Evolence/Lidocaine: Assess injection pain of Evolence/Lidocaine
  collagen: Injectable collagen
  Lidocaine: admix anesthetic
Arm/Group | Pain Assessment for Evolence/Topical Anesthetic | Pain Assessment for Evolence/Lidocaine
Number analyzed (Participants) | 10 | 10
Number analyzed (nasolabial folds) | 10 | 10
units on a scale | 5.2 (2.1) | 2.0 (0.8)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Pain Assessment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No